CLINICAL TRIAL: NCT04166305
Title: Clinical and Genetic Factors Associated With Drug Resistance of Epilepsy
Brief Title: Drug Resistant Epilepsy: Clinical and Genetic Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University Hospital 6
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Epilepsy, Drug Resistant
Keywords: Epilepsy, genetic and drug resistant
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Drug responders: 60 patients are drug responders
  Interventions: Genetic: Genetic study for SCN1A c.3184 A/G and CCL2-2518G>A polymorphism:
- Drug resistant: 60 patients are drug resistant
  Interventions: Genetic: Genetic study for SCN1A c.3184 A/G and CCL2-2518G>A polymorphism:
- The control: The control consists of 60 Age and gender matched healthy individual with negative past and family history of epilepsy and febrile convulsion.
  Interventions: Genetic: Genetic study for SCN1A c.3184 A/G and CCL2-2518G>A polymorphism:

INTERVENTIONS:
Genetic: Genetic study for SCN1A c.3184 A/G and CCL2-2518G>A polymorphism: — DNA analysis: Genomic DNA will be extracted from EDTA-anticoagulated peripheral blood (QIAamp DNA Blood mini kit,QIAGEN).
  Genotyping of SCN1A c.3184 A/G(rs2298771) polymorphism

SUMMARY:
This study is to identify the clinical criteria of drug resistant epilepsy and to explore whether SCN1A c.3184 A/G (rs2298771) and ccl2(rs1024611) polymorphisms could serve as genetic based biomarkers to predict drug resistance among epileptic patient.

DETAILED DESCRIPTION:
This retrospective case control study will be conducted on 120 epileptic patients treated with AEDs, 60 patients are drug responders and 60 patients are drug resistant. All epileptic patient will be recruited from outpatient epilepsy clinic, Department of Neurology, Mansoura University hospital. The control consists of 60 Age and gender matched healthy individual with negative past and family history of epilepsy and febrile convulsion.

Subjects:

Inclusion criteria:

1. Patient with diagnosis of epilepsy (idiopathic or cryptogenic/symptomatic), according to the International League Against Epilepsy classification confirmed by electroencephalogram.
2. Treatment with at least one AED, long enough to achieve the optimal dose; drug-resistance and drug-responsiveness, according to the criteria ILAE 2010.
3. Written consent obtained from a patient or legal guardian.

Exclusion criteria:

1. Patient with severe adverse anti epileptic drug reactions.
2. Patient with unreliable records of seizure frequency.
3. Patient with poor compliance with AEDs,.
4. Patient with significant psychiatric comor- bidity,
5. Patient with progressive systemic disorders .
6. Patient with history of alcohol or drug abuse.
7. Epileptic patients in clinical remission or with gradual withdrawal of therapy.
8. Epileptic patients with therapy titration phase.

Methods:

After an informed consent, all participants will be subjected to the following;

1. A detailed history taking; including age, sex, age of onset , type of seizure, duration of epilepsy, pretreatment and post treatment seizure frequency , and drugs (antiepileptic drugs, others).
2. Full laboratory investigation including (complete blood count, liver function test, serum creatinine, electrolyte assay, thyroid profile, blood sugar test).
3. Serum level of antiepileptic drug.
4. Electroencephalogram in order to localize site of paroxysmal activity.
5. MRI brain: T1, T2 and FLAIR: axial and coronal cuts to detect any structural abnormalities,
6. Both control and epileptic patient will underwent genetic study for SCN1A c.3184 A/G and CCL2-2518G>A polymorphism:

   * DNA analysis:

Genomic DNA will be extracted from EDTA-anticoagulated peripheral blood (QIAamp DNA Blood mini kit,QIAGEN).

ELIGIBILITY:
Inclusion Criteria:

* Patient with diagnosis of epilepsy (idiopathic or cryptogenic/symptomatic), according to the International League Against Epilepsy classification confirmed by electroencephalogram.
* Treatment with at least one AED, long enough to achieve the optimal dose; drug-resistance and drug-responsiveness, according to the criteria ILAE 2010.

Exclusion Criteria:

* Patient with severe adverse anti-epileptic drug reactions.
* Patient with unreliable records of seizure frequency.
* Patient with poor compliance with AEDs,.
* Patient with significant psychiatric comorbidity,
* Patient with progressive systemic disorders .
* Patient with history of alcohol or drug abuse.
* Epileptic patients in clinical remission or with gradual withdrawal of therapy.
* Epileptic patients with therapy titration phase.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This retrospective case control study will be conducted on 120 epileptic patients treated with AEDs, 60 patients are drug responders and 60 patients are drug resistant. The control consists of 60 Age and gender matched healthy individual with negative past and family history of epilepsy and febrile convulsion.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Genetic study for SCN1A c.3184 A/G and CCL2-2518G>A polymorphism: | 5-7 days
  • DNA analysis: Genomic DNA will be extracted from EDTA-anticoagulated peripheral blood (QIAamp DNA Blood mini kit,QIAGEN).
  • Genotyping of SCN1A c.3184 A/G(rs2298771) polymorphism

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] He X, Li Y, Liu Z, Yue X, Zhao P, Hu J, Wu G, Mao B, Sun D, Zhang H, Song X, Wang Y, Shao J. The association between CCL2 polymorphisms and drug-resistant epilepsy in Chinese children. Epileptic Disord. 2013 Sep;15(3):272-7. doi: 10.1684/epd.2013.0603. PMID 23996681
- [Result] Kumari R, Lakhan R, Garg RK, Kalita J, Misra UK, Mittal B. Pharmacogenomic association study on the role of drug metabolizing, drug transporters and drug target gene polymorphisms in drug-resistant epilepsy in a north Indian population. Indian J Hum Genet. 2011 May;17 Suppl 1(Suppl 1):S32-40. doi: 10.4103/0971-6866.80357. PMID 21747585
- [Result] Kasperaviciute D, Sisodiya SM. Epilepsy pharmacogenetics. Pharmacogenomics. 2009 May;10(5):817-36. doi: 10.2217/pgs.09.34. PMID 19450130
- [Result] Kwan P, Arzimanoglou A, Berg AT, Brodie MJ, Allen Hauser W, Mathern G, Moshe SL, Perucca E, Wiebe S, French J. Definition of drug resistant epilepsy: consensus proposal by the ad hoc Task Force of the ILAE Commission on Therapeutic Strategies. Epilepsia. 2010 Jun;51(6):1069-77. doi: 10.1111/j.1528-1167.2009.02397.x. Epub 2009 Nov 3. PMID 19889013
- [Result] Lakhan R, Kumari R, Misra UK, Kalita J, Pradhan S, Mittal B. Differential role of sodium channels SCN1A and SCN2A gene polymorphisms with epilepsy and multiple drug resistance in the north Indian population. Br J Clin Pharmacol. 2009 Aug;68(2):214-20. doi: 10.1111/j.1365-2125.2009.03437.x. PMID 19694741
- [Result] Lorigados Pedre L, Morales Chacon LM, Orozco Suarez S, Pavon Fuentes N, Estupinan Diaz B, Serrano Sanchez T, Garcia Maeso I, Rocha Arrieta L. Inflammatory mediators in epilepsy. Curr Pharm Des. 2013;19(38):6766-72. doi: 10.2174/1381612811319380009. PMID 23530510
- [Result] Manna I, Gambardella A, Bianchi A, Striano P, Tozzi R, Aguglia U, Beccaria F, Benna P, Campostrini R, Canevini MP, Condino F, Durisotti C, Elia M, Giallonardo AT, Iudice A, Labate A, La Neve A, Michelucci R, Muscas GC, Paravidino R, Zaccara G, Zucca C, Zara F, Perucca E. A functional polymorphism in the SCN1A gene does not influence antiepileptic drug responsiveness in Italian patients with focal epilepsy. Epilepsia. 2011 May;52(5):e40-4. doi: 10.1111/j.1528-1167.2011.03097.x. PMID 21561445
- [Result] Marchi N, Granata T, Freri E, Ciusani E, Ragona F, Puvenna V, Teng Q, Alexopolous A, Janigro D. Efficacy of anti-inflammatory therapy in a model of acute seizures and in a population of pediatric drug resistant epileptics. PLoS One. 2011 Mar 28;6(3):e18200. doi: 10.1371/journal.pone.0018200. PMID 21464890
- [Result] Pohlmann-Eden B, Weaver DF. The puzzle(s) of pharmacoresistant epilepsy. Epilepsia. 2013 May;54 Suppl 2:1-4. doi: 10.1111/epi.12174. PMID 23646961
- [Result] Sanchez MB, Herranz JL, Leno C, Arteaga R, Oterino A, Valdizan EM, Nicolas JM, Adin J, Armijo JA. Genetic factors associated with drug-resistance of epilepsy: relevance of stratification by patient age and aetiology of epilepsy. Seizure. 2010 Mar;19(2):93-101. doi: 10.1016/j.seizure.2009.12.004. Epub 2010 Jan 12. PMID 20064729
- [Result] Tellez-Zenteno JF, Hernandez-Ronquillo L, Buckley S, Zahagun R, Rizvi S. A validation of the new definition of drug-resistant epilepsy by the International League Against Epilepsy. Epilepsia. 2014 Jun;55(6):829-34. doi: 10.1111/epi.12633. Epub 2014 May 14. PMID 24828683
- [Result] Wirrell EC. Predicting pharmacoresistance in pediatric epilepsy. Epilepsia. 2013 May;54 Suppl 2:19-22. doi: 10.1111/epi.12179. PMID 23646966
- [Result] Walker L, Sills GJ. Inflammation and epilepsy: the foundations for a new therapeutic approach in epilepsy? Epilepsy Curr. 2012 Jan;12(1):8-12. doi: 10.5698/1535-7511-12.1.8. PMID 22368518